CLINICAL TRIAL: NCT04151225
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled, Repeat Dose, Dose-ranging Phase 2a/2b Study to Evaluate the Safety, Tolerability and Efficacy of an Anti-oncostatin M Monoclonal Antibody (GSK2330811) in Patients With Moderate to Severe Crohn's Disease
Brief Title: Study to Evaluate Safety, Tolerability and Efficacy of GSK2330811 in Crohn's Disease
Acronym: COSMIS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Internal sponsor decision to terminate project in Crohn's disease due to potential narrow therapeutic window. No subjects were enrolled
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 208482
Record Dates: First submitted 2019-11-04; First posted 2019-11-05 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Crohns Disease; Crohn's Disease
Keywords: Monoclonal antibody; Crohns Disease; Oncostatin M; GSK2330811
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: This is a parallel group treatment study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double blind study where participants, investigator and sponsor will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Participants receiving placebo (Placebo Comparator): Participants will receive placebo loading dose followed by placebo for 12 weeks during Induction phase. Participants with clinical response at Week 12 will continue to receive placebo into a 40-weeks blinded maintenance period. Participants without a clinical response at Week 12 will receive a 450mg GSK2330811 SC loading dose at Week 12, followed by 150 mg SC every week from Week 13 until Week 23, followed by 150 mg SC every 2 weeks until Week 50.
  Interventions: Drug: Placebo
- Participants receiving GSK2330811 450mg loading dose/150mg Q1W (Experimental): Participants will receive 450mg GSK2330811 SC as loading dose followed by 150 mg GSK2330811 Q1W for 12 weeks during Induction period. Participants with clinical response at Week 12 will continue into a 40 weeks blinded maintenance period will receive 150 mg GSK2330811 SC Q2W. Participants without a clinical response will receive GSK2330811 150mg Q1W from Week 12 until Week 23, followed by GSK2330811 150mg Q2W until Week 50.
  Interventions: Drug: GSK2330811
- Participants receiving GSK2330811 300mg loading dose/150mg Q2W (Experimental): Participants will receive 300mg GSK2330811 SC as loading dose followed by 150mg GSK2330811 SC Q2W for 12 weeks during Induction period. Participants with clinical response at Week 12 will continue into a 40 weeks blinded maintenance period will receive 150mg GSK2330811 SC Q2W. Participants without a clinical response will receive GSK2330811 150mg Q1W from Week 12 until Week 23, followed by GSK2330811 150mg Q2W until Week 50.
  Interventions: Drug: GSK2330811
- Participants receiving GSK2330811 300mg loading dose/150mg Q4W (Experimental): Participants will receive 300mg GSK2330811 SC as loading dose followed by 150mg GSK2330811 SC Q4W for 12 weeks during Induction period. Participants with clinical response at Week 12 will continue into a 40 weeks blinded maintenance period will receive 150 mg GSK2330811 SC Q4W. Participants without a clinical response will receive GSK2330811 150mg Q1W from Week 12 until Week 23, followed by GSK2330811 150mg Q2W until Week 50.
  Interventions: Drug: GSK2330811
- Participants receiving GSK2330811 150mg Q8W (Experimental): Participants will receive GSK2330811 SC 150 mg Q8W for 12 weeks during Induction period. Participants with clinical response at Week 12 will continue into a 40 weeks blinded maintenance period will receive 150 mg GSK2330811 SC Q8W. Participants without a clinical response will receive GSK2330811 150mg Q1W from Week 12 until Week 23, followed by GSK2330811 150mg Q2W until Week 50.
  Interventions: Drug: GSK2330811

INTERVENTIONS:
Drug: GSK2330811 — GSK2330811 will be available as SC injection with a unit dose strength of 150 mg/mL. GSK2330811 will be available in single-use pre-filled syringe.
  Arms: Participants receiving GSK2330811 150mg Q8W; Participants receiving GSK2330811 300mg loading dose/150mg Q2W; Participants receiving GSK2330811 300mg loading dose/150mg Q4W; Participants receiving GSK2330811 450mg loading dose/150mg Q1W
Drug: Placebo — Placebo will be available as SC injection of 0.9 percent saline solution. It will be available as single-use pre-filled syringe.
  Arms: Participants receiving placebo

SUMMARY:
The study will include participants with moderate to severe Crohn's disease. The aim is to evaluate the safety, tolerability, and efficacy of anti-oncostatin M monoclonal antibody (mAb) GSK2330811. This is a parallel group study with Induction and Maintenance periods. During Induction, the first 100 participants randomised will receive a 450mg GSK2330811 SC loading dose followed by 150mg weekly (Q1W), or placebo for 12 weeks. Additional dose-ranging arms will open after the 100th participant is randomized and in addition to placebo and the highest dose arms will also include a 300mg subcutaneous (SC) loading dose followed by 150mg SC every 2 weeks (Q2W) arm, a 300mg loading dose followed by 150mg SC every 4 weeks (Q4W) arm and a 150mg SC every 8 weeks (Q8W) arm. Participants with a clinical response at Week 12 will continue into a 40-week blinded maintenance period and will receive either 150mg SC Q2W, 150mg SC Q4W, 150mg SC Q8W or placebo. Participants without a clinical response at Week 12 will be offered up to 40 weeks of open label treatment with GSK2330811. Approximately 560 participants will be screened to randomize 280.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 years of age or over at the time of signing the informed consent.
* Participants who have a diagnosis of Crohn's Disease, established at least 3 months prior to first screening visit, supported by radiologic, histologic and/or endoscopic findings, and are expected to be able to be managed on an outpatient basis, if clinical course does not worsen.
* Participants who have active colitis and/or ileitis at screening, confirmed by centrally-read ileo-colonoscopy, defined as a baseline SES-CD score of >= 7 (>= 4 if disease confined to the terminal ileum) and <=35.
* Participants who have active clinical disease at Baseline, measured by PRO2, defined as a 7-day average SF >= 4 and/or a 7-day average AP >=2.
* Participants who have a history of at least one of the following: Inadequate response to, loss of response to, or intolerance to conventional immunosuppression (i.e. azathioprine, 6-mercaptopurine, methotrexate); Inadequate response to, loss of response to, intolerance to, or demonstrated dependence on oral corticosteroids; Inadequate response to, loss of response to, or intolerance to biologic therapy or small molecule JAK inhibitors.
* Participants with Baseline body mass index (BMI) >= 18.5 kilogram per square meter (kg/m^2).
* Male and Female participants are both eligible to participate.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: Not a woman of childbearing potential (WOCBP) or A WOCBP who agrees to use a contraceptive method that is highly effective, with a failure rate of <1 percent, from 28 days prior to first dosing day (Day 1), during the dosing period and for at least 126 days (18 weeks) after the last dose of study treatment, corresponding to the time needed to eliminate any study intervention. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.
* Participant who is capable of giving signed informed consent.

Exclusion Criteria:

* Participants with a current diagnosis of indeterminate colitis, inflammatory bowel disease (unclassified), infectious colitis, lymphocytic colitis, microscopic colitis, radiation colitis, ischemic colitis or ulcerative colitis.
* Participants with complications of Crohn's disease including strictures, adhesions, stenosis, short bowel syndrome and any other manifestation, if it is anticipated to require surgery during the study or that could interfere with study assessments (including but not limited to symptomatic strictures or stenosis) or that may confound the evaluation of benefit from treatment with GSK2330811.
* A current ileostomy or colostomy.
* Any bowel resection or diversion within 6 months or other intra-abdominal surgery within 3 months prior to the screening ileo-colonoscopy.
* Receiving tube feeding, defined formula diets, or total parenteral nutrition within 4 weeks prior to the screening ileo-colonoscopy.
* Current or prior abscess (proven or suspected) unless drained and adequately treated at least 3 weeks prior to the screening ileo-colonoscopy for cutaneous and perianal abscesses and at least 8 weeks prior to the screening ileo-colonoscopy for intra-abdominal abscesses. There must be no anticipated need for further surgery during the study.
* Active fistulas associated with an abscess and anticipated need for surgery during the study. If a fistula is present, it should have established drainage.
* Prior fecal micro-biota transplant within 3 months prior to the screening ileo-colonoscopy.
* Participants with any uncontrolled medical conditions, other than active Crohn's Disease, that in the opinion of the investigator puts the participant at unacceptable risk or likely will interfere with study assessments or data integrity. Other medical conditions should be stable at the time of screening expected to remain stable for the duration of the study.
* Known history of or current bleeding or coagulation disorder.
* Current or chronic history of liver or biliary disease (except for Gilbert's syndrome, asymptomatic gallstones or uncomplicated fatty liver disease).
* A major organ transplant (example heart, lung, kidney, liver, pancreas) or hematopoietic stem cell/marrow transplant.
* Unstable lifestyle factors, such as alcohol use to excess or recreational drug use, to the extent that in the opinion of the investigator would interfere with the ability of a participant to complete the study.
* Major surgery within 3 months prior to the first screening visit or planned during the study.
* Cancer or carcinoma in situ present within the last 5 years, except for adequately treated non-metastatic basal or squamous cell cancers of the skin or carcinoma in situ of the uterine cervix that has been fully treated and shows no evidence of recurrence.
* Active infection, or a history of infection as follows: Active or unresolved infection (i.e. bacterial, viral, fungal or parasitic). This does not include minor localized infections such as fungal nail infections, at the investigator's discretion; Infection requiring treatment with antimicrobials (i.e. antibacterial, antiviral, anti-parasitic or antifungal agents), where the last dose of antimicrobials falls within 4 weeks prior to the screening ileo-colonoscopy. This does not include topical antimicrobials, which are permitted; History of opportunistic infection (example Cytomegalovirus [CMV] colitis, disseminated herpes zoster), that has not resolved within 6 months prior to the screening ileo-colonoscopy or of recurrent infections, as determined by the investigator. This does not include infections that may occur in immunocompetent individuals, such as fungal nail infections or vaginal candidiasis, unless of an unusual severity or frequency.
* Evidence of active or latent tuberculosis (TB) as documented by medical history and examination, and TB testing: either a positive tuberculin skin test (TST; defined as a skin induration >5 millimeter [mm] at 48 to 72 hours, regardless of Bacillus Calmette-Guerin [BCG] or other vaccination history) or a positive (not indeterminate) QuantiFERON-TB Gold test; Positive Clostridium difficile toxin test during screening. However, rescreening can be undertaken following documented successful treatment.
* Symptomatic herpes zoster within 3 months prior to the screening ileo-colonoscopy.
* Intravenous, intramuscular or rectal corticosteroids within 2 weeks prior to the screening ileo-colonoscopy.
* Oral corticosteroids at a dose greater than 20mg/day prednisolone (or equivalent) within 2 weeks prior to the screening ileo-colonoscopy. A dose <= 20mg/day is permitted but this must have been at a stable dose for 2 weeks prior to the screening ileo-colonoscopy and participant and investigator assesses that the participant is likely able to maintain this stable dose until the Week 12 visit.
* Budesonide at a dose greater than 6mg/day within 2 weeks prior to the screening ileocolonoscopy. A dose <= 6mg/day is permitted but this must have been at a stable dose for 2 weeks prior to the screening ileo-colonoscopy and participant and investigator should be willing to maintain this stable dose until the Week 12 visit.
* Any anti-Tumour necrosis factor (TNF) biologic within 8 weeks prior to screening ileo-colonoscopy and/or detectable blood levels within 8 weeks following last anti- TNF dose.
* Vedolizumab within 8 weeks prior to screening ileo-colonoscopy.
* Ustekinumab within 8 weeks prior to screening ileo-colonoscopy.
* Rituximab within 1 year prior to screening ileo-colonoscopy.
* Any previous treatment with alemtuzumab or natalizumab.
* Other biologic therapies/ or novel targeted therapies used for the treatment of Crohn's disease not mentioned in this section, unless approved by the Medical Monitor.
* Treatment with interferon, thalidomide, or methotrexate within 8 weeks prior to the screening ileo-colonoscopy, or treatment with methotrexate within 4 weeks prior to the screening ileo-colonoscopy.
* Treatment with azathioprine and 6-mercaptopurine unless on a stable dose for 8 weeks prior to the screening ileo-colonoscopy and participant and investigator should be willing to maintain this stable dose until the end of the follow-up period.
* Treatment with 5-aminosalicylates and sulfasalazine unless on a stable dose for 4 weeks prior to the screening ileo-colonoscopy and participant and investigator should be willing to maintain this stable dose until the end of the follow-up period.
* Live vaccine(s) within 4 weeks prior to the screening ileo-colonoscopy or plans to receive such vaccines during the study.
* Treatment with full dose anti-coagulant medications, including warfarin, heparin, thrombin inhibitors, and Factor Xa inhibitors within 2 weeks prior to the screening ileo-colonoscopy.
* Treatment with anti-platelet medications (example clopidogrel, prasugrel, ticagrelor and dipyridamole) within 2 weeks prior to the screening ileo-colonoscopy. This does not include aspirin at doses of 150 mg or less, or non-steroidal anti-inflammatory drugs, which are permitted.
* Receipt of an investigational product as part of participation in an interventional clinical trial within the following time period, prior to the Day 1 visit: 3 months, 5 half-lives, or twice the duration of the biological effect of the investigational product.
* Prior exposure to GSK2330811.
* Diagnostic assessments at screening: Hemoglobin < 110 grams per Liter (g/L); Platelet count < 150*10^9/L; Presence of Hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to first dose of study treatment; Presence of the Hepatitis B core antibody (HBcAb) even if HBsAg is negative; Positive Hepatitis C antibody test result at screening or within 3 months prior first dose of study treatment; Positive Hepatitis C Ribonucleic acid (RNA) test results at screening or within 3 months prior to first dose of study treatment; Positive human immunodeficiency virus (HIV) antibody test; Estimated glomerular filtration rate Modification of Diet in Renal Disease (MDRD) calculation of <45 milliliter (mL) per minute per 1.73m^2; Alanine transferase (ALT) > 2 times upper limit of normal (ULN); Bilirubin > 1.5 times ULN (isolated bilirubin > 1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* QT corrected (QTc) >450 millisecond (msec) or QTc >480msec for participants with bundle branch block. The QTc is the QT interval corrected for heart rate according to Bazett's formula (QTcB), Fridericia's formula (QTcF) or another method, either machine-read or manually over-read. The same correction formula should be used throughout the study.
* Where participation in the study would result in the donation of in excess of 500 mL blood over a 3-month period.
* Clinically significant multiple or severe drug allergies (including to humanized monoclonal antibodies), known hypersensitivity to GSK2330811 or any excipients used in the clinical formulation of GSK2330811, intolerance to topical corticosteroids, or a history of severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A [IgA] dermatosis, toxic epidermal necrolysis and exfoliative dermatitis).
* Any other history of significant allergy that in the opinion of the investigator contraindicates their participation in this study.
* Participants who, in the opinion of the investigator, would be unable to complete the daily diaries independently example unable to read and/or understand the questions being asked.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-05 (Estimated); Primary Completion 2024-04-22 (Estimated); Study Completion 2025-05-26 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with endoscopic response measured by Simple Endoscopic score for Crohn's Disease (SES-CD) at Week 12 | Week 12
  The SES-CD is a validated tool for grading the endoscopic severity of active Crohn's disease based on an assessment of the size of individual ulcers, the proportion of the surface that is abnormal and the proportion of the surface that is ulcerated, and the presence or absence of visible stenosis. The attributes are scored across 5 bowel segments and combined to give an SES-CD score ranging from 0 to 56 (higher scores represent more severe endoscopic disease involvement). SES-CD will be determined for each endoscopy using a central reading algorithm. Endoscopic response is defined as >= 50 percent decrease from Baseline in SES-CD

SECONDARY OUTCOMES:
Percentage of participants with endoscopic response based on dose response relationship at Week 12 measured by SES-CD | Week 12
  The SES-CD is a validated tool for grading the endoscopic severity of active Crohn's disease based on an assessment of the size of individual ulcers, the proportion of the surface that is abnormal and the proportion of the surface that is ulcerated, and the presence or absence of visible stenosis. The attributes are scored across 5 bowel segments and combined to give an SES-CD score ranging from 0 to 56 (higher scores represent more severe endoscopic disease involvement). SES-CD will be determined for each endoscopy using a central reading algorithm. Endoscopic response is equivalent to >= 50 percent decrease from Baseline in SES-CD
Change from Baseline in SES-CD at Week 12 | Baseline (within 35 days prior to Day 1) and Week 12
  The SES-CD is a validated tool for grading the endoscopic severity of active Crohn's disease based on an assessment of the size individual ulcers, the proportion of the surface that is abnormal and the proportion of the surface that is ulcerated, and the presence or absence of visible stenosis. The attributes are scored across 5 bowel segments and combined to give an SES-CD score ranging from 0 to 56 (higher scores represent more severe endoscopic disease involvement). SES-CD will be determined for each endoscopy using a central reading algorithm
Percentage of participants in endoscopic remission at Week 12 | Week 12
  Endoscopic remission will be equivalent to SES-CD <=4 and >=2 point reduction from Baseline, and no sub-score > 1 in any individual score
Percentage of participants with absence of mucosal ulceration on endoscopy at Week 12 | Week 12
  Endoscopy mucosal healing will be assessed during central endoscopic reading of the ileo-colonoscopies where absence of mucosal ulceration will be noted
Percentage of participants with clinical response measured by Patient Reported Outcome 2 (PRO2) at Week 12 | Week 12
  Participants will record the following items related to patient reported symptoms/outcomes information electronically on a hand-held device at home during the study: Abdominal pain (AP) in the past 24 hours (scored from 0 to 3: 0 = none, 1 = mild, 2 = moderate and 3 = severe); Number of liquid or very soft stools (stool frequency; SF) in the past 24 hours. Clinical response will be defined as >=30 percent reduction from Baseline in average daily SF or >=30 percent reduction from Baseline in average daily AP, with both not worse than Baseline.
Percentage of participants in clinical remission at Week 12 measured by PRO2 | Week 12
  Participants will record the following items related to patient reported symptoms/outcomes information electronically on a hand-held device at home during the study: Abdominal pain (AP) in the past 24 hours (scored from 0 to 3: 0 = none, 1 = mild, 2 = moderate and 3 = severe); Number of liquid or very soft stools (stool frequency; SF) in the past 24 hours. Clinical remission is defined as average daily SF <=3 and average daily AP <=1, with both not worse than Baseline
Change from Baseline in serum C-reactive protein at Week 12 | Baseline (Day 1) and Week 12
  Serum samples will be collected at indicated timepoints for the analysis of changes from Baseline of C-reactive protein.
Change from Baseline in fecal calprotectin at Week 12 | Baseline (Day 1) and Week 12
  Change from Baseline of fecal calprotectin will be assessed by collecting fecal samples at the time-points
Plasma concentration of GSK2330811 | Pre-dose on Day 1 and Weeks 1, 2, 3, 4, 6, 8, 10, and 12
  Blood samples will be collected at indicated timepoints for analysis of plasma concentration of GSK2330811
Area Under the Concentration Time Curve Over the Dosing Period (AUC [0-tau]) of GSK2330811 | Pre-dose on Day 1 and Weeks 1, 2, 3, 4, 6, 8, 10, and 12
  Blood samples will be collected at indicated timepoints for analysis of AUC (0-tau) of GSK2330811
Trough Concentration at steady state (Ctrough ss) | Pre-dose on Day 1 and Weeks 1, 2, 3, 4, 6, 8, 10, and 12
  Blood samples will be collected at indicated time-points for analysis of Ctrough ss of GSK2330811
Serum levels of free Oncostatin M (OSM) | Pre-dose on Day 1 and Weeks 1, 2, 3, 4, 6, 8, 10, and 12
  Blood samples will be collected at indicated timepoints for analysis of free OSM levels in serum.
Serum levels of total OSM | Pre-dose on Day 1 and Weeks 1, 2, 3, 4, 6, 8, 10, and 12
  Blood samples will be collected at indicated timepoints for analysis of total OSM levels in serum.
Number of participants with anti-drug antibodies | Pre-dose on Day 1 and Weeks 4, 8 and 12
  Blood samples will be collected at indicated timepoints for analysis of anti-drug antibodies

OTHER OUTCOMES:
Number of participants with serious adverse events (SAEs) | Up to Week 68
  A SAE is defined as any untoward medical occurrence that at any dose may result in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly or birth defect and important medical events may jeopardize the participants or may require medical or surgical intervention to prevent one of the other outcomes listed above.
Number of participants with adverse events (AEs) and Adverse Event of Special Interest (AESI) | From Week 0 (Day 1) to Week 68
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Complications of Anemia, Complications of Thrombocytopenia, Injection site reactions like rash, allergic reaction and infusion like reactions; Hypersensitivities like anaphylaxis and angioedema; Opportunistic Infections and Delayed wound healing will be considered as AESI.
Number of participants with clinically significant changes in systolic blood pressure (SBP) and diastolic blood pressure (DBP) | Week 0 (Day 1) to Week 68
  SBP and DBP will be measured in a semi-supine position after 5 minutes rest.
Number of participants with clinically significant changes in temperature | Week 0 (Day 1) to Week 68
  Temperature will be measured in a semi-supine position after 5 minutes rest.
Number of participants with clinically significant changes in pulse rate | Week 0 (Day 1) to Week 68
  Pulse rate will be measured in a semi-supine position after 5 minutes rest.
Number of participants with clinically significant changes in hematology parameters | Week 0 (Day 1) to Week 68
  Clinically significant abnormal laboratory findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Laboratory assessment for hematology parameters will include platelet count, hemoglobin, red blood cell (RBC) count, hematocrit, Red cell distribution width, mean corpuscular volume (MCV), percentage reticulocytes, mean corpuscular hemoglobin concentration (MCHC) and mean corpuscular hemoglobin (MCH). White blood cell (WBC) count with differential will include neutrophils, lymphocytes, monocytes, eosinophil and basophils. Additional hematology parameters included serum ferritin, percentage transferrin saturation, iron, serum B12, serum folate, and serum haptoglobin.
Number of participants with clinically significant changes in clinical chemistry parameters | Week 0 (Day 1) to Week 68
  Clinically significant abnormal laboratory findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Laboratory assessment for clinical chemistry parameters will include blood urea nitrogen (BUN), potassium, calcium, sodium, creatinine, glucose, total cholesterol, triglycerides, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, C-reactive protein, total protein, albumin, total and direct bilirubin, lactate dehydrogenase, estimated glomerular filtration rate, high density lipoprotein and low density lipoprotein.
Number of participants with clinically significant changes in urinalysis | Week 0 (Day 1) to Week 68
  Clinically significant abnormal laboratory findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Laboratory assessment for urinalysis parameters will include specific gravity, concentration of hydrogen ions (pH), glucose, protein, blood, ketones, bilirubin, nitrite, leukocytes by dipstick, microscopic examination if blood, protein or leukocytes are abnormal.
Number of participants with clinically significant changes in 12- lead Electrocardiogram (ECG) | From Screening visit (within 35 days prior to Day 1) to Week 68
  Triplicate 12-lead ECGs will be obtained using an ECG machine, that automatically measures PR, QRS, QT and Corrected QT (QTc) intervals.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com